CLINICAL TRIAL: NCT06456554
Title: Acellular Dermal Matrix Investigation in Breast Reconstruction
Acronym: ADMIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI Surgical (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTI-CL-5000
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acellular Dermal Matrix (Experimental): Breast reconstruction with Cortiva Tissue Matrix
  Interventions: Device: Acellular Dermal Matrix (Cortiva Tissue Matrix)
- no Acellular Dermal Matrix (No Intervention): Breast reconstruction only with no ADM

INTERVENTIONS:
Device: Acellular Dermal Matrix (Cortiva Tissue Matrix) — non-crosslinked dermis
  Arms: Acellular Dermal Matrix

SUMMARY:
Prospective, multi-center, dual-arm non-randomized clinical study in females undergoing a two-stage breast reconstruction using a pre-pectoral technique.

ELIGIBILITY:
Inclusion Criteria:

* Genetic female
* Age 22 or older at time of consent
* Undergoing immediate breast reconstruction
* 2 stage breast reconstruction using pre pectoral technique
* Nipple or skin sparing mastectomy
* Willing and capable of providing informed consent
* Able to comply with study requirements

Exclusion Criteria:

* Planned concurrent reconstruction with pedicled flaps or free tissue
* Pregnant or breast feeding
* Investigator has determined tissue is unsuitable for two-stage breast reconstruction
* History of psychological characteristics that may be incompatible with the surgical procedure and the prosthesis
* Any serious and/or unstable pre-existing medical disorder or other conditions that could interfere with the subject's safety, the informed consent process, or compliance with the study protocol, in the opinion of the investigator
* Vulnerable subject populations
* Currently participating in another clinical trial that would have the potential to interfere or conflict with the treatment, follow-up, or objectives of this study
* Prior history of neoadjuvant radiotherapy to the reconstruction site or chest wall
* Active abscess or infection in the intended reconstruction site
* Residual gross tumor at the intended reconstruction site
* Active use of any tobacco/nicotine products
* Has body mass index (BMI) >35
* Uncontrolled diabetes defined as HbA1c ≥7 within 3 months prior to stage 1 procedure
* Is currently taking medications including systemic steroids

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse events | 12 months
  Surgery-related adverse events requiring rehospitalization or reoperation of the breast under study
Health related quality of life | 12 months
  Change from baseline in quality of life as measured by the BREAST-Q Physical Well-Being

SECONDARY OUTCOMES:
Change in quality of life | 1 year and 2 years
  Change from baseline in quality of life as measured by the BREAST-Q
Procedure related adverse events | 3 months, 1 year and 2 years
  Rate of procedure-related adverse events requiring additional treatment
Investigational device related adverse events | 3 months, 1 year and 2 years
  Rate of investigational device-related adverse events requiring additional treatment
Histopathology assessment | stage 2 procedure
  Histopathology assessment at stage 2 procedure

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Arkansas, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado, Aurora, Colorado
  - Washington University, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Mercy Hospital, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No